CLINICAL TRIAL: NCT06701929
Title: How Fasting Duration Before Cesarean Section Affects the Quality of Recovery Score (ObsQoR-11)
Brief Title: The Impact of Fasting Duration on Quality of Recovery After Cesarean Section
Status: Recruiting | Type: Observational
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Matthew Cameron, MDCM MPH, Associate Professor, Jewish General Hospital
Other Study IDs: ObsQoR-11 Survey (2025-4422)
Record Dates: First submitted 2024-11-20; First posted 2024-11-22 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Quality Improvement; Quality of Recovery From Anaesthesia; Cesarean Section; Fasting ( 6H for Solid ; 2H for Clear Fluid )
Keywords: Quality of Recovery; cesarean section; fasting duration
MeSH Terms: conditions — Fasting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will evaluate the effect of fasting duration and elective c-section start time on the overall quality of recovery. Patients will be seen 24 hours after surgery to answer 11 questions on their overall recovery after surgery. Several factors will be tracked to determine their effect on recovery, with the primary variable of interesting

DETAILED DESCRIPTION:
This is a prospective observational study aiming to evaluate the impact of fasting time before cesarean section on the quality of recovery after c-section. All patients presenting for elective cesarean section with low transverse incision, under spinal anesthesia will be considered for inclusion.

The primary outcome will be the ObsQoR-11 score approximately 24 hours after surgery. Secondary outcomes will include the presence of nausea, vomiting or retching during surgery, the volume of intravenous fluid administered, the dose of vasopressor administered, the pain scores two hours after surgery, and the dose of opioid used in the 24 hours after surgery.

The primary analysis will be a linear regression to determine if there is a statistically significant correlation between fasting time and the ObsQoR-11 score while factoring in the variables mentioned above. Secondary analyses will determine if the fasting duration correlates with a change in any of the eleven components of the ObsQoR-11 score or the secondary outcomes listed. In addition, the fasting data will be plotted against the ObsQoR-11 score to determine if an inflection point is present.

Ten observations will be obtained for each independent variable included in the model, for a total of 100 patients in the study.

ELIGIBILITY:
Inclusion Criteria:

* Presenting for elective c-section under spinal anesthesia

Exclusion Criteria:

* Unable to communicate in French or English
* Urgent c-section
* Planned general anesthesia

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients presenting to the Jewish General Hospital for elective cesarean section under spinal anesthesia will be considered for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2025-03-18 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Obstetric Quality of Recovery (ObsQoR-11) | 3 months
  Obstetric quality of recovery after c-section, which has been validated based on the total score of 11 questions, with total scores ranging from 0 to 110, where 0 is the worst, and 110 is the best.

SECONDARY OUTCOMES:
Nausea & Vomitting | 24 hours
  The presence of nausea vomiting or retching during or within 24 hours of surgery
Numeric Rating Scale (NRS) Pain Score 2 hours after surgery | 2 hours after surgery
  Rating of pain, on a scale where 0 is no pain, and 10 is the worst pain imaginable.

CONTACTS AND LOCATIONS:
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data
Supporting Information: Study Protocol, SAP
Time Frame: After publication for two years

REFERENCES:
- [Background] Kielty J, Borkowska A, Lawlor E, El-Khuffash AF, Doherty A, O'Flaherty D. Use of the Obstetric Quality-of-Recovery score (ObsQoR-11) to measure the impact of an enhanced recovery programme for elective caesarean section. Int J Obstet Anesth. 2024 Feb;57:103955. doi: 10.1016/j.ijoa.2023.103955. Epub 2023 Nov 10. PMID 38030526
- [Background] Bollag L, Lim G, Sultan P, Habib AS, Landau R, Zakowski M, Tiouririne M, Bhambhani S, Carvalho B. Society for Obstetric Anesthesia and Perinatology: Consensus Statement and Recommendations for Enhanced Recovery After Cesarean. Anesth Analg. 2021 May 1;132(5):1362-1377. doi: 10.1213/ANE.0000000000005257. PMID 33177330
- [Background] Ciechanowicz S, Setty T, Robson E, Sathasivam C, Chazapis M, Dick J, Carvalho B, Sultan P. Development and evaluation of an obstetric quality-of-recovery score (ObsQoR-11) after elective Caesarean delivery. Br J Anaesth. 2019 Jan;122(1):69-78. doi: 10.1016/j.bja.2018.06.011. Epub 2018 Jul 31. PMID 30579408